CLINICAL TRIAL: NCT07363070
Title: Adherence to Chronic Positive Airway Pressure Therapy in Obese Patients With Sleep-disordered Breathing
Status: Completed | Type: Observational
Sponsor: Anne Kathrine Staehr-Rye (Other)
Responsible Party: Sponsor-Investigator, Anne Kathrine Staehr-Rye, Associate professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: p-2025-20420
Record Dates: First submitted 2026-01-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disorder; Breathing-Related; Obesity; Adherence, Treatment
MeSH Terms: conditions — Sleep Wake Disorders; Obesity; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Positive Airway Pressure Therapy — Use of Positive Airway Pressure Therapy
Device: Positive Airway Pressure Therapy — Use of chronic positive Airway Pressure Therapy

SUMMARY:
To describe the adherence to positive airway pressure therapy among obese adult patients refered to the respiratory center east

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Body mass index above 30 kg/m2
* Referred to the Respiratory Center East between january 2021 and january 2024

Exclusion Criteria:

* Neuromuscular disease
* Spinal cord injury
* Craniofacial malformation
* Scoliosis
* Diaphragmatic paresis
* Referred to profylactic secrete management only
* Already in treatment with nPAP with use of nPAP a minimum of 4 hours per night for 70% of the time within a consecutive 30-day period during the last 90 days.
* No medical indication for start of nPAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respiratory center east,
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Compliance to noninvasive positive airway pressure therapy (nPAP) - 90 days | 0-3 months after start of noninvasive positive airway pressure therapy
  Use of nPAP a minimum of 4 hours per night for 70% of the time within a consecutive 30-day period within the first 90 days of having the equipment.

SECONDARY OUTCOMES:
Mortality | 1 year
  Mortality up to 1 year after initiation of noninvasive positive airway pressure therapy
Compliance to noninvasive positive airway pressure therapy (nPAP) - 1 year | Time Frame: 275 to 365 day after start of noninvasive positive airway pressure therapy
  Use of nPAP a minimum of 4 hours per night for 70% of the time within a consecutive 30-day period within the 275 to 365 day of having the equipment.

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Center East, Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided